CLINICAL TRIAL: NCT06062849
Title: Is it Really Necessary to Insert a Nephrostomy Tube or Double J Stent in Percutaneous Nephrolithotomy?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bursa City Hospital (Other Government)
Responsible Party: Principal Investigator, abdullah erdogan, associate professor, Bursa City Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-KAEK-140 / 2023-12/2
Record Dates: First submitted 2023-09-13; First posted 2023-10-02 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Kidney Calculi; Postoperative Pain
Keywords: percutaneous nephrolithotomy; nephrostomy tube; double J stent
MeSH Terms: conditions — Kidney Calculi; Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- totally tubeless (Active Comparator): there is no nephrostomy tube or double J (JJ) stent
  Interventions: Procedure: totally tubless
- tubeless (Active Comparator): only JJ stent
  Interventions: Device: double J stent
- nephrostomy tube (Experimental): nephrostomy tube
  Interventions: Device: nephrostomy tube

INTERVENTIONS:
Device: nephrostomy tube — we will investigate if a nephrostomy tube really necessary after PNL operations
  Arms: nephrostomy tube
Device: double J stent — we will investigate if a JJ stent really necessary after PNL operations
  Arms: tubeless
Procedure: totally tubless — we will not insert any device after the procedure and investigate if a nephrostomy tube or JJ stent really necessary after PNL operations
  Other Names: there is no device
  Arms: totally tubeless

SUMMARY:
In this study, investigators aimed to compare the postoperative pain status and comfort situations depending on instruments used in the percutaneous nephrolithotomy operation

DETAILED DESCRIPTION:
A total of 90 patients aged 18 and over will undergo percutaneous nephrolithotomy (PNL) for kidney stones of 2 cm or more between 01/08/2023 and 01/02/2024 will be included in the study. Preoperative demographic data of the patients, body mass index (BMI), stone size and stone location, hemogram, biochemistry, coagulation parameters, urine analysis, and urine culture test results will be recorded. Radiological evaluation will be obtained according to computerized tomography (CT) data. While patients aged 18 years and above with kidney stones larger than 2 cm were included in the study, patients under 18 years of age, patients with anatomical anomalies (horseshoe kidney, ectopic kidney, ureteropelvic junction stenosis, ureteral stenosis), patients with uncorrectable bleeding diathesis, bilateral kidney stones will not be included in the study.

Patients who do not have major complications (serious bleeding, renal pelvis perforation) after the PNL procedure and residual stones cannot be detected according to the scopic image obtained will be randomized and divided into three groups. Patients in the first group will not be fitted with a Double J (JJ) stent and/or nephrostomy (Completely Tubeless), patients in the second group will only be fitted with a JJ stent, and patients in the third group will only be fitted with a 14 French Malecot nephrostomy. The patients' pain scores, analgesic use, hemoglobin values, operation success, complications, and additional procedure requirements in the postoperative period will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and above
* Larger than 2 cm kidney stones

Exclusion Criteria:

* Under 18 years of age
* Anatomical anomalies (horseshoe kidney, ectopic kidney, ureteropelvic junction stenosis, ureteral stenosis),
* Uncorrectable bleeding diathesis
* Bilateral kidney stones

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
postoperative pain | 6 months
  investigators will compare postoperative pain status between the three groups with a Visual Analog Scale (VAS) questionnaire at 0, 1, 6, 12, and 24 hours postoperatively. Participants will rate their pain on a scale of 1 to 10 in ascending order.
postoperative urine leakage | 6 months
  Researchers will investigate whether there is a difference in urine leakage between the three groups by measuring the number of pads changed daily.

CONTACTS AND LOCATIONS:
Overall Officials: Sedat Oner, MD, Study Director — Bursa City Hospital
Locations (1):
- Bursa City Hospital, Bursa, Turkey (Türkiye)